CLINICAL TRIAL: NCT02918838
Title: Supporting Adolescents to Adhere - an Intervention Using Airtime Rewards Allocated by a Prize Drawing
Acronym: SATA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAND (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3R01HD074925-04S1 (NIH)
Record Dates: First submitted 2016-09-14; First posted 2016-09-29 (Estimated); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Human Immunodeficiency Virus
Keywords: HIV; Antiretroviral (ARV); co-trimoxazole; SMS; Lottery incentive; mobile health; Uganda; Youth
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Own Adherence Group (Experimental): Participant chooses their adherence level to be reached at next clinic visit (at least 80%, but can be higher). If they reach that percentage measured using the MEMS cap, they can participate in a lottery for an airtime reward of none, a small amount, and a larger amount. Participants also receive a weekly motivational message reminding them of their incentive to adhere. If they respond to the message they will receive airtime top-up.
  Interventions: Behavioral: Own Adherence Group
- Fixed Adherence Group (Experimental): Participant is told to meet a pre-determined target of 90%. If they reach that percentage measured using the MEMS cap, they can participate in a lottery for an airtime reward of none, a small amount, and a larger amount. Participants also receive a weekly motivational message reminding them of their incentive to adhere. If they respond to the message they will receive airtime top-up.
  Interventions: Behavioral: Fixed Adherence Group
- Control Group (Active Comparator): Participants do not receive a lottery incentive conditional on adherence. Participants will however, continue to receive weekly messaging with airtime top-up contingent on response.
  Interventions: Behavioral: Control Group

INTERVENTIONS:
Behavioral: Own Adherence Group — Participant chooses their adherence level to be reached at next clinic visit (at least 80%, but can be higher). If they reach that percentage measured using the MEMS cap, they can participate in a lottery for an airtime reward of none, a small amount, and a larger amount. Participants also receive a weekly motivational message reminding them of their incentive to adhere. If they respond to the message they will receive airtime top-up.
  Arms: Own Adherence Group
Behavioral: Fixed Adherence Group — Participant is told to meet a pre-determined target of 90%. If they reach that percentage measured using the MEMS cap, they can participate in a lottery for an airtime reward of none, a small amount, and a larger amount. Participants also receive a weekly motivational message reminding them of their incentive to adhere. If they respond to the message they will receive airtime top-up.
  Arms: Fixed Adherence Group
Behavioral: Control Group
  Arms: Control Group

SUMMARY:
This study is an extension of Reminding Adolescents to Adhere (RATA) (Unique protocol ID: 1R01HD074925-01). Participants for SATA will be recruited during the RATA month 24 exit survey.

Participants will be randomized 1:1:1 into either one of two intervention group (receiving the weekly messages and a chance to draw a prize at each clinic visit based on either a fixed adherence level of 90% or a self-chosen one of at least 80% as further detailed below) or the control group that receives the existing RATA intervention consisting of weekly motivational messages and the chance to get mobile airtime rewards conditional on responding. Doing so will allow the investigators to cleanly evaluate the impact of these additional adherence-based lotteries, and guarantees that those who have been in the control group receiving standard of care in the first 24 months of the RATA intervention will also receive an intervention for reasons of fairness.

DETAILED DESCRIPTION:
* For Group 1 (lottery reward with fixed target): Study coordinators check participant's MEMS extraction for last month's adherence. Study coordinators then tell participants of the participants' adherence in the last month. Participants are also informed that during the next clinic visit, if they adhere at least 90 percent they have a chance to enter into a game where they have a chance of winning mobile airtime, by drawing into a bag and picking a card associated with their airtime winnings. If they do not have 90% adherence, they will not receive the airtime award game, but there will be another chance the next time they come for their scheduled clinic visit during the study period.
* For Group 2 (lottery award with own target): Study coordinators check participant's MEMS extraction for last month's adherence. They inform participants of their adherence in the last month. In order to be eligible for an airtime reward game, during their next clinic visit they must reach their own target goal. The target adherence goal must be greater than 80%. Participants may, for example, choose 80%, 85%, 90%, 95%, or 100%. Again, if they meet or exceed this target they have a chance to draw into a bag to win mobile airtime. If they do not have meet this self-imposed target adherence, they will not be eligible to play the airtime award game, but there will be another chance the next time they come for their scheduled clinic visit during the study period.

During each clinic visit, participants will have their MEMS extracted and study coordinators will check for average adherence between that day and the last clinic visit. For those who have met the target, coordinators will initiate the lottery, complete the drawing procedure, or send them the airtime reward without drawing (depending on which group).

Every Sunday, study investigators will send treatment participants a motivational message to remind them about the reward. Within each of the two intervention groups, study investigators will randomly send the message either in a loss-frame or a gain-frame, i.e. an intervention participant (in either group) will some weeks receive a message telling them to keep up motivation (as a code-word for adherence) to win a prize, and some weeks telling them to make sure not to lose their chance to win a prize.

ELIGIBILITY:
Inclusion Criteria:

* have been in HIV care at the clinic for at least three months
* are currently taking HIV-related medication (ART or co-trimoxazole)
* either own a phone or have regular access to one
* intend to stay at the clinic for the study period
* are not in boarding school (where phones are forbidden)

Exclusion Criteria:

- does not speak or understand either English or Luganda

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 216 (Actual)
Dates: Start 2016-08; Primary Completion 2018-02-01 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
Medication adherence rates using electronically monitored adherence (MEMS cap) data | 9 months after enrollment
  Medication Event Monitoring System (MEMS)-cap data will be collected continuously over the course of the 9-month study period allowing the study investigators to investigate daily adherence and its timing. MEMS caps data indicating the date and time when the participant opened their pill bottle (either one of the ART medications or prophylaxis if not on ART yet) will be used to calculate the primary outcome variable of adherence (# of actual bottle openings / # of prescribed bottle openings).

SECONDARY OUTCOMES:
Fraction of clients displaying adherence of 90% or more | 9 months after enrollment
  MEMS caps data indicating the date and time when the participant opened their pill bottle (either one of the ART medications or prophylaxis if not on ART yet) will be used to calculate the secondary outcome measures of fraction of clients displaying adherence of 90% or more.
Indicator for treatment interruptions of more than 48 hours | 9 months after enrollment
  MEMS caps data indicating the date and time when the participant opened their pill bottle (either one of the ART medications or prophylaxis if not on ART yet) will be used to calculate the secondary outcome measures of an indicator for treatment interruptions of more than 48 hours.
Viral load assays | 9 months after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Linnemayr, PhD, Principal Investigator — RAND
Locations (1):
- Mildmay Uganda, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: Undecided